CLINICAL TRIAL: NCT02137616
Title: Effectiveness of Antipsychotic Drugs to Treat Psychosis Syndrome: an Open Label, Controlled Study
Brief Title: Antipsychotic to Treat Psychosis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, xiaofeng Guo, prof., Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201002003
Record Dates: First submitted 2014-05-05; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Psychotic Disorders
Keywords: psychosis; syndrome; risk; antipsychotic
MeSH Terms: conditions — Psychotic Disorders; Syndrome | interventions — Risperidone; Olanzapine; Quetiapine Fumarate; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- risperidone (Active Comparator): low dosage of antipsychotic drug
  Interventions: Drug: risperidone
- olanzapine (Active Comparator): low doseage of antipsychotic
  Interventions: Drug: olanzapine
- quetiapine (Active Comparator): low doseage of antipsychotic
  Interventions: Drug: Quetiapine
- aripiprazole (Active Comparator): low doseage of antipsychotic
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: risperidone — Risperdal tablets
  Other Names: Risperidol
  Arms: risperidone
Drug: olanzapine — olanzapine tablets
  Other Names: olanzapine tablets
  Arms: olanzapine
Drug: Quetiapine — quetiapine tablets
  Other Names: quetiapine tablets
  Arms: quetiapine
Drug: Aripiprazole — Aripiprazole tablets
  Other Names: Aripiprazole tablets
  Arms: aripiprazole

SUMMARY:
This study assess the safety and effects of atypical antipsychotics in subjects with psychosis syndrome and psychosis risk syndrome.

DETAILED DESCRIPTION:
The investigators investigated whether administration of atypical antipsychotics could alleviate prodromal symptoms and be well tolerated by subjects with psychosis syndrome and psychosis risk syndrome.

ELIGIBILITY:
Inclusion Criteria:

* were help-seeking young individuals in outpatients service
* aged 16-30 years
* fitted one of the following Criteria: Psychosis-risk Syndromes (COPS-SIPS) or Psychotic Syndrome (POPS-SIPS) or DSM-IV diagnosis of schizophreniform disorder

Exclusion Criteria:

* a previous diagnosis of any psychotic disorder or bipolar disorders according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition;
* symptoms fully accounted for by an Axis 1 disorder or sequelae of drug/alcohol use;
* neurological disorders or organic disorders affecting the central nervous system, substance-related disorders or mental retardation as defined by the DSM-IV criteria;
* history treatment of antipsychotic or antidepression, mood stabilizers or electroconvulsive therapy;
* diagnosed as having a serious and unstable medical condition.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Changes of PANSS total scores from baseline to 18 months | 18 months

SECONDARY OUTCOMES:
Social function | 18 months
  Social function was assessed by the Global Assessment of Functioning (GAF) every three month
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 18 months
  Adverse Events were assessed at baseline and every month after treatments

CONTACTS AND LOCATIONS:
Overall Officials: xiaofeng Guo, Dr, Principal Investigator — the second xiangya hospitcal
Locations (1):
- the Second Xiangya Hospital, Changsha, Hunan, China